CLINICAL TRIAL: NCT01777256
Title: An Adaptive Phase II Study to Evaluate the Efficacy, Pharmacodynamics, Safety and Tolerability of GSK2586184 in Patients With Mild to Moderate Systemic Lupus Erythematosus
Brief Title: An Adaptive Phase II Study to Evaluate the Efficacy, Pharmacodynamics, Safety and Tolerability of GSK2586184
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study met a protocol defined futility criterion and will be terminated following completion of the Follow Up Visit on the last subject randomised.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115919
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; adaptive design; clinical safety and efficacy; pharmacodynamics
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — GSK2586184

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- GSK2586184 50 mg Arm (Experimental): Subjects in the GSK2586184 50 mg Arm will receive twice daily dose of GSK2586184 50 mg 1 x 50 mg tablet + 1x placebo tablet) orally up to 12 weeks. Study medication should be taken with food, immediately following a meal
  Interventions: Drug: GSK2586184 50 mg; Drug: Placebo
- GSK2586184 100 mg Arm (Experimental): Subjects in the GSK2586184 100 mg Arm will receive twice daily dose of GSK2586184 100 mg (2 x 50 mg tablets) orally up to 12 weeks. Study medication should be taken with food, immediately following a meal.
  Interventions: Drug: GSK2586184 100 mg
- GSK2586184 200 mg Arm (Experimental): Subjects in the GSK2586184 200 mg Arm will receive twice daily dose of GSK2586184 200 mg (1 x 200 mg tablet + 1x placebo tablet) orally up to 12 weeks. Study medication should be taken with food, immediately following a meal.
  Interventions: Drug: GSK2586184 200 mg; Drug: Placebo
- GSK2586184 400 mg Arm (Experimental): Subjects in the GSK2586184 400 mg Arm will receive twice daily dose of GSK2586184 400 mg (2 x 200 mg tablets) orally up to 12 weeks. Study medication should be taken with food, immediately following a meal.
  Interventions: Drug: GSK2586184 400 mg
- Placebo (Placebo Comparator): Subjects in the placebo arm will receive twice daily dose of 2 matching placebo tablets orally up to 12 weeks; taken with food, immediately following a meal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2586184 50 mg — GSK2586184 tablet will be administered orally as twice daily dose of 50 mg (1 x 50 mg tablet) up to 12 weeks.
  Arms: GSK2586184 50 mg Arm
Drug: GSK2586184 100 mg — GSK2586184 tablet will be administered orally as twice daily dose of (2 X 50 mg tablet) up to 12 weeks.
  Arms: GSK2586184 100 mg Arm
Drug: GSK2586184 200 mg — GSK2586184 tablet will be administered orally as twice daily dose of 200 mg (1 x 200 mg) up to 12 weeks.
  Arms: GSK2586184 200 mg Arm
Drug: GSK2586184 400 mg — GSK2586184 tablet will be administered orally as twice daily dose of (2 X 200 mg) up to 12 weeks.
  Arms: GSK2586184 400 mg Arm
Drug: Placebo — Matching placebo tablet will be administered orally twice daily up to 12 weeks.
  Arms: GSK2586184 200 mg Arm; GSK2586184 50 mg Arm; Placebo

SUMMARY:
This is an adaptive, dose ranging, Phase II study to investigate the relationship between repeat doses of GSK2586184 and the pharmacodynamic effect and clinical efficacy in patients with active systemic lupus erythematosus (SLE). This study will also investigate the safety and tolerability of repeat doses of GSK2586184. During the study, up to 3 Interim Analyses will be conducted. These are to monitor the pharmacodynamic effect and safety following 2 weeks of therapy (Interim Analysis 1); and the clinical efficacy and safety of GSK2586184 following 12 weeks of therapy (Interim Analyses 2 and 3). Subjects who meet the entry criteria (approximately 150 to 250) will be randomized in a 1:1:1:1:1 ratio to receive GSK2586184 at doses of 50 milligram (mg) twice daily (b.i.d), 100 mg b.i.d, 200 mg b.i.d, 400 mg b.i.d or Placebo b.i.d. GSK2586184 tablets available in 50 and 200 mg dose strength will be administered orally up to 12 weeks.

Subjects who complete the study will participate in the study for approximately 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age & Gender: Male or female between 18 and 75 years of age inclusive
* SLE classification: a clinical diagnosis of SLE according to the American College of Rheumatology (ACR) classification criteria
* Severity of disease: clinically active SLE disease defined as a SELENA SLEDAI score ≥8 at screening
* Auto antibodies: serologically active having unequivocally positive anti-nuclear antibody (ANA) or anti-double stranded DNA (anti-dsDNA) antibody test results from 2 independent time points
* Treatment for SLE: patient stable on either no treatment or a stable dose of: corticosteroids (<=15 mg/day prednisolone or equivalent) and /or hydroxychloroquine (<=400 mg daily dose) Subjects receiving azathioprine (<=2 mg/kg/day or <=150 mg/day, whichever is greater) or mycophenolate mofetil (<=1.5 g/day), or methotrexate (MTX) (<=20 mg/week), either alone or in addition to steroids and / or hydroxychloroquine
* Prevention of Pregnancy:

A female Subject is eligible to participate if she is not pregnant or nursing; is of non-childbearing potential. Females of child-bearing potential must agree to use one highly effective contraception method in addition to barrier protection OR two forms of highly effective contraception.

* Informed consent: Capable of giving written informed consent

Exclusion Criteria:

* Kidney Disease: meeting any of the following criteria:

Proteinuria > 0.5g/24 hour OR equivalent spot urine protein to creatinine ratio of 0.5mg/mg; Serum creatinine > 1.5 X upper limit of normal (ULN); active nephritis requiring acute therapy not permitted by protocol; required peritoneal dialysis or hemodialysis or high dose corticosteroid (> 100 mg/day prednisone or equivalent) within 90 days prior to first dose; active renal disease shown on renal biopsy in the three months prior to screening.

* CNS Disease: active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident [CVA], cerebritis or CNS vasculitis) requiring therapeutic intervention within 60 days prior to first dose.
* Alcohol Abuse: Evidence or, in the opinion of the investigator, suspicion of alcohol consumption exceeding national guidelines and / or symptoms of alcohol dependency.
* Substance abuse: evidence of current recreational drug abuse or dependence.
* Hepatitis B: A positive pre-study Hepatitis B surface antigen or anti-Hepatitis B core antibody test at screening
* Hepatitis C: A positive Hepatitis C antibody at screening.
* HIV: A positive test for HIV antibody
* Previous Investigational Product Exposure:

The subject has participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) prior to the first dosing day in the current study; OR exposure to more than four new chemical entities within 12 months prior to the first dosing day.

* Previous and current medication: Use of prescription or non-prescription drugs, including: agents known to interact with GSK2586184, erythopoetic stimulation factors; vitamins, herbal and dietary supplements
* Prior biological therapies: treatment with a biological therapy within the last 12 months
* Transplantation: Have a history of a major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Uncontrolled Other Diseases: Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to SLE which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk.
* Surgery and Other Conditions: Have a planned surgical procedure or a history of any other medical disease laboratory abnormality, or condition that, in the opinion of the investigator, makes the subject unsuitable for the study.
* Cancer: Have a history of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.-
* Infections: have required management of acute or chronic infections as follows: currently on any suppressive therapy for a chronic infection (such as pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria); OR hospitalisation for treatment of infection OR use of parenteral (IV or intramuscular) antibiotics (antibacterials, antivirals, anti-fungals, or anti parasitic agents) within 60 days prior to first dose.
* Mycobacterium Tuberculosis: Known latent or active infection with Mycobacterium Tuberculosis. Screening procedures consistent with local guidelines should be implemented.
* Haematology: neutrophil count <=1.5 X 10^9/L, Hb <=10g/dL, lymphocyte count <=350/mm^3 or 0.35 x 10^9/L and platelet count <=100 X 10^9/L
* Serum immunoglobulin (Ig) levels: IgG and/or IgM <= the lower limit of normal (LLN)
* Liver function tests: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >=2x upper limit of normal (ULN); alkaline phosphatase and bilirubin >1.5xULN (isolated bilirubin >1.5ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Other laboratory abnormalities: Any Grade 3 or 4 haematology or clinical chemistry laboratory abnormality
* Drug sensitivity: History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Blood donation: Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-03-01; Primary Completion 2014-03-01 (Actual); Study Completion 2014-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage Inhibition from Baseline of interferon (IFN) Transcriptional Biomarkers at Week 2 | Baseline(Day1) and Week 2
  Mean reduction (40%) from Baseline of the IFN transcriptional signature biomarker was monitored at Week 2. Percentage (Per) inhibition (=[(Day x-Baseline)/Baseline]*-100), was the Per reduction from Baseline (Day1) and evaluated in any pre-designated panels of genes i.e. Addenbrookes 1, Addenbrookes 2, JAK439, PD, Panel Stripping, Flare and Transcription. Analysis was performed using a repeated measures model with covariates of treatment, baseline, Day, Day by baseline and Day by treatment interactions. Only those Par available at the specified time points were analysed (n=X,X,X,X,X). Different Par may have been analysed at different time points, so the overall number of Par analysed reflects everyone in the Intent To Treat (ITT) Population i.e. Par randomised to treatment, received >=1 dose of study medication and had >=1 valid post dose assessment
Change from Baseline of SELENA SLEDAI score at indicated time points up to Week 16 | Baseline(Day1), Weeks 2, 4, 6, 8, 10, 12 and 16
  The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) is a validated index for assessing SLE disease activity. It is a weighted index in which signs and symptoms, laboratory tests, and physician's assessment for each of 9 organ systems are given a weighted score and summed, if present at the time of the visit or in the preceding 10 days. Modified version of SLEDAI is Safety of Estrogen in Lupus National Assessment (SELENA) SLEDAI where the maximum theoretical score for the SELENA SLEDAI was 105 with 0 indicating inactive disease. Baseline value is defined as Day 1 (pre-dose) SELENA SLEDAI score.
Change from Baseline in systolic blood pressure and diastolic blood pressure at the indicated time points up to Week 16 | Baseline(Day1), Weeks 2, 4, 6, 8, 10, 12 and 16
  Change from Baseline in systolic blood pressure (BP) and diastolic BP is summarized for each post-Baseline assessment up to Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in heart rate at the indicated time points up to Week 16 | Baseline (Day 1), Weeks 2, 4, 6, 8, 10, 12 and 16
  Change from Baseline in sitting and supine heart rate is summarized for each post-Baseline assessment up to Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last pre-treatment value observed.
Change from Baseline in temperature at the indicated time points up to Week 16 | Baseline (Day 1), Weeks 2, 4, 6, 8, 10, 12 and 16
  Change from Baseline in temperature is summarized for each post-Baseline assessment up to Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in albumin, globulin and protein at the indicated time points up to Week 16 | Baseline (Day 1), Weeks 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the albumin, globulin and protein values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from baseline in alkaline phosphatase, alanine amino transferase, aspartate amino transferase, creatine kinase, gamma glutamyl transferase and lactate dehydrogenase at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the alkaline phosphatase (ALP), alanine amino transferase (ALT), aspartate amino transferase (AST), creatine kinase (CK), gamma glutamyl transferase (GGT) and lactate dehydrogenase (LDH) values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in anion gap, calcium, cholesterol, chloride, carbon dioxide, glucose, HDL cholesterol, potassium, LDL cholesterol, magnesium, phosphate, soidium, triglycerides, urea, VLDL cholesterol at the indicated time points up to Week 16 | Baseline (Day 1), Weeks 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the anion gap, calcium, ionised calcium, cholesterol, chloride, carbon dioxide, glucose, high density lipoprotein (HDL) cholesterol (fasted and not fasted), potassium, low density lipoprotein (LDL) cholesterol (fasted and not fasted), magnesium, phosphate, sodium, triglycerides (fasted and not fasted), urea and very low density lipoprotein (VLDL) cholesterol values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in bilirubin, creatinine, iron binding capacity, iron and urate at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the bilirubin, direct and indirect bilirubin, creatinine, total iron binding capacity (TIBC), unsaturated iron binding capacity (UIBC), iron and uric acid values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in albumin/globulin, BUN/creatinine and transferrin saturation at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from baseline in the albumin/globulin, blood urea nitrogen (BUN)/creatinine and transferrin saturation values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in creatinine clearance at the indicated time points up to Week 16 | Baseline (Day 1), Weeks 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the Creatinine Clearance values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in basophils, eosinophils, lymphocytes, monocytes, neutrophils, neutrophils segmented (SG), platelets and leukocytes at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 1, 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the basophils, eosinophils, lymphocytes, monocytes, neutrophils, neutrophils segmented (SG), platelets and leukocytes values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in basophils/leukocytes, eosinophils/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes, neutrophils/leukocytes, neutrophils SG/leukocytes and erythrocyte distribution width (EDW) at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 1, 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the basophils/leukocytes, eosinophils/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes, neutrophils/leukocytes, neutrophils segmented (SG)/leukocytes and erythrocyte distribution width (EDW) values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in erythrocytes and reticulocytes at the indicated time points up to Week 16 | Baseline (Day 1), Weeks 1, 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the erythrocyte and reticulocyte values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in hemoglobin and erythrocyte mean corpuscular hemoglobin concentration (EMCHC) at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 1, 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the hemoglobin and erythrocyte mean corpuscular hemoglobin concentration (EMCHC) values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in erythrocyte mean corpuscular hemoglobin (EMCH) at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 1, 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the hemoglobin and erythrocyte mean corpuscular hemoglobin (EMCH) values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in erythrocyte mean corpuscular volume (EMCV) and mean platelet volume (MPV) at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 1, 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the erythrocyte mean corpuscular volume (EMCV) and mean platelet volume (MPV) values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in hematocrit and reticulocytes/erythrocytes at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 1, 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the hematocrit and reticulocytes/erythrocytes values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Number of participants with urinalysis data at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 1, 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Number of participants with negative and positives (trace, +, ++ and +++) data for urine glucose (UGLU), urine ketones (UKET) and urine occult blood (UOB) are summarized for each post-Baseline assessment until Week 16. Urinalysis was performed by dipstick method. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in urine protein at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the urine protein values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Change from Baseline in urine protein/creatinine at the indicated time points up to Week 16 | Baseline(Day 1), Weeks 2, 3, 4, 5, 6, 8, 10, 12 and 16
  Change from Baseline in the urine protein/creatinine values are summarized for each post-Baseline assessment until Week 16. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Number of participants with any adverse events (AEs) and any serious adverse events (SAEs) up to Week 16 | Up to Week 16
  An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign(including an abnormal laboratory finding), symptom, or disease(new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, a congenital anomaly/birth defect, important medical events that jeopardize the participants or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition.
Number of participants with severity Grade 1, 2, 3, 4 and 5 adverse events (AEs) | Up to 16 Weeks
  The Common Terminology Criteria for Adverse Events (CTCAE, Version 4) has categorised AEs in five grades. Grade refers to the severity of the AE. Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.

SECONDARY OUTCOMES:
SRI Response Rate at Week 4, 8, 12 and 16 | Week 4, 8, 12 and 16
  The relationship between dose of GSK2586184 and clinical response was assessed by the SLE Responder Index (SRI). The percentage of participants achieving a response on the composite endpoint are summarized. Response is defined as:>= 4 point reduction from the Baseline in the SELENA SLEDAI score and no worsening (increase of <0.30 points from the Baseline) in Physicians Global Assessment (PGA),and no new British Isles Lupus Assessment Group (BILAG) A organ domain score or 2 new BILAG B organ domain scores compared with the Baseline. Baseline value is defined as the last Pre-treatment value observed.
Change from baseline in SLEDAI-2K score and the S2K RI-50 score over time (up to Week 12) | Baseline(Day 1) to Week 12
  The relationship between dose of GSK2586184 and clinical response was assessed by Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) and SLEDAI-2K Responder Index 50 (S2K RI-50) scores. SLEDAI-2K is a revised version of the SLEDAI in which the persistent active disease in the items rash, alopecia, mucosal ulcers and proteinuria would be scored as opposed to new occurrences as are measured in the SLEDAI. S2K RI-50 detects a minimum 50% improvement in disease manifestations among lupus participants. It covers 9 organ systems, utilising the same 24 descriptors and reflects disease activity over the previous 30 days. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed. Due to early termination of the study, data for this endpoint was not summarized.
Mean GSK2586184 plasma concentrations on Weeks 2, 4, 6, 8, 10 and 12 | Weeks 2, 4, 6, 8, 10 and 12
  Plasma pharmacokinetic (PK) pre-dose (PRD) samples were collected for all participants at Weeks 2, 4, 8, 10 and 12 prior to the morning dose. At Week 2, additional blood sample were collected at 1hour (hr) and 4 hr post-dose (POD) and at Week 6, additional blood sample were collected, from 6 hr to 10 hr POD. PK Population comprised of all participants randomised to treatment, who have taken at least one dose. Only participants for whom plasma PK samples were obtained were assessed (represented by n=X,X,X,X in category titles). Different participants may have been analysed at different time points, so the overall number of participants analysed reflects everyone in the Pharmacokinetic(PK) Population.
Area under the concentration-time curve over the dosing interval (AUC[0-tau]) up to Week 12 | Weeks 2, 4, 6, 8, 10 and 12
  Plasma PK PRD samples were collected for all participants at Weeks 2, 4, 8, 10 and 12 prior to the morning dose. At Week 2, additional blood sample were collected at 1hr and 4 hr POD and at Week 6, additional blood sample were collected, from 6 hr to 10 hr POD. AUC(0-tau).is calculated from a population pharmacokinetic model using Non Linear Mixed Effect Model (NONMEM) after log-transformation of PK data. Only participants for whom plasma PK samples were obtained and assessed.
Apparent clearance (CL/F) up to Week 12 | Weeks 2, 4, 6, 8, 10 and 12
  Plasma PK PRD samples were collected for all participants at Weeks 2, 4, 8, 10 and 12 prior to the morning dose. At Week 2, additional blood sample were collected at 1hr and 4 hr POD and at Week 6, additional blood sample were collected, from 6 hr to 10 hr POD. CL/F is calculated, as dose divided by AUC(0-tau), from a population pharmacokinetic model using Non Linear Mixed Effect Model (NONMEM) after log-transformation of PK data. Only participants for whom plasma PK samples were obtained and assessed.
Volume of distribution (Vss) up to Week 12 | Weeks 2, 4, 6, 8, 10 and 12
  Plasma PK PRD samples were collected for all participants at Weeks 2, 4, 8, 10 and 12 prior to the morning dose. At Week 2, additional blood sample were collected at 1hr and 4 hr POD and at Week 6, additional blood sample were collected, from 6 hr to 10 hr POD. Apparent volume of distribution is calculated as dose divided by (AUC[0-tau] lambda z) where lambda z is the terminal phase rate constant. Vss is calculated from a population pharmacokinetic model using Non Linear Mixed Effect Model (NONMEM) after log-transformation of PK data. Only participants for whom plasma PK samples were obtained and assessed
Mean change from Baseline in the SF-36 Domain Scores up to Week 16 | Baseline(Day 1), Weeks 12 and 16
  The Short Form (36) Health Survey (SF-36v2 ) is a participant-reported survey of participant health and measures general health-related quality of life. There are 36 items grouped into nine health domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, Mental Health, Reported health transition (RHT). SF-36v2 gives a score for each of these domains based on the questions as assessed by participants. The lower the score the more disability and the higher the score the less disability. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Mean change from Baseline in the Brief Fatigue Inventory (BFI) Domain Score up to Week 16 | Baseline (Day 1), Weeks 2, 4, 6, 8, 10, 12 and 16
  The BFI was developed to quickly measure severity of fatigue in participants as well as its impact on their ability to function over the previous 24 hrs. It consists of nine items that look at fatigue in the past that are rated on a 0 -10 numeric rating scale where 0 is no fatigue or does not interfere and 10 is bad fatigue or completely interferes with activity. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.
Mean change from Baseline in the Brief Pain Inventory (BPI) Domain Score up to Week 16 | Baseline(Day 1), Weeks 2, 4, 6, 8, 10, 12 and 16
  The BPI is a questionnaire used to assess the severity of pain and the impact of pain on daily functioning in the following areas: general activity, mood, walking ability, normal work, including outside the home and housework, relations with other people, enjoyment of life and sleep. Two sub scores are derived from questionnaire: the worst pain score and the interference score. To derive a valid worst pain score, a minimum of 3 (out of 6) non missing values were required versus 4 (out of 7) for the interference score. Change from Baseline was calculated as the individual post-Baseline value minus the Baseline value. Baseline value is defined as the last Pre-treatment value observed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (47):
- Argentina (3):
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, San Juan
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- Czechia (2):
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- GSK Investigational Site, Tallinn, Estonia
- France (5):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
- Germany (5):
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Herne, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Jena, Thuringia
- Greece (4):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion-Crete
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Thessaloniki
- Hong Kong (3):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin
  - GSK Investigational Site, Tuenmen
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Zalaegerszeg
- Peru (4):
  - GSK Investigational Site, La Victoria, Lima region
  - GSK Investigational Site, San Borja, Lima region
  - GSK Investigational Site, Surco, Lima region
  - GSK Investigational Site, Lima
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Poznan
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
- South Africa (4):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Parow
  - GSK Investigational Site, Pinelands, Cape Town
  - GSK Investigational Site, Stellenbosch
- GSK Investigational Site, Seoul, South Korea
- Spain (3):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Linköping

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kahl L, Patel J, Layton M, Binks M, Hicks K, Leon G, Hachulla E, Machado D, Staumont-Salle D, Dickson M, Condreay L, Schifano L, Zamuner S, van Vollenhoven RF; JAK115919 Study Team. Safety, tolerability, efficacy and pharmacodynamics of the selective JAK1 inhibitor GSK2586184 in patients with systemic lupus erythematosus. Lupus. 2016 Nov;25(13):1420-1430. doi: 10.1177/0961203316640910. Epub 2016 Jul 11. PMID 27055521
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 115919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115919 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register